CLINICAL TRIAL: NCT07287098
Title: preEMBER: A Phase 2, Open-label Study Evaluating Imlunestrant in Premenopausal Women With Estrogen Receptor-Positive, HER2-Negative Breast Cancer
Brief Title: A Study of Imlunestrant (LY3484356) in Premenopausal Women With Estrogen Receptor-Positive (ER+) Human Epidermal Growth Factor Receptor 2 Negative (HER2-) Early Breast Cancer
Acronym: PreEMBER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27511; 2025-523258-15-00 (EU CTIS Number); J2J-MC-JZLL (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-12-11; First posted 2025-12-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Breast Neoplasm Female
MeSH Terms: interventions — Imlunestrant; Goserelin; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Imlunestrant (Active Comparator): Imlunestrant will be given orally
  Interventions: Drug: Imlunestrant
- Imlunestrant + Goserelin (Active Comparator): Imlunestrant will be given orally and Goserelin will be given Subcutaneously (SC)
  Interventions: Drug: Imlunestrant + Goserelin; Device: pre-filled syringe
- Tamoxifen (Active Comparator): Tamoxifen will be given orally
  Interventions: Drug: Tamoxifen 20 mg

INTERVENTIONS:
Drug: Imlunestrant — Given Orally
  Other Names: LY3484356
  Arms: Imlunestrant
Drug: Imlunestrant + Goserelin — Imlunestrant will be given orally and Goserelin will be administered SC
  Other Names: LY3484356
  Arms: Imlunestrant + Goserelin
Drug: Tamoxifen 20 mg — Given Orally
  Arms: Tamoxifen
Device: pre-filled syringe — SC
  Arms: Imlunestrant + Goserelin

SUMMARY:
This study will include two groups of patients: Cohort 1 and Cohort 2.

Cohort 1: will help researchers learn how a medicine called imlunestrant (LY3484356) affects a specific type of breast cancer. Some patients will take both imlunestrant and another treatment to suppress their ovarian function. Some will take it without ovarian suppression. Researchers will compare the effects in breast cancer cells to those of another medicine called tamoxifen. All patients in this group will be premenopausal women who have a type of early breast cancer called estrogen receptor-positive, HER2-negative. The treatment in this group will last for up to 29 days.

Cohort 2: will help researchers understand how imlunestrant affects the ovaries when it is taken without ovarian suppression. This group will also include premenopausal women with the same type of breast cancer. The treatment in this group will last for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

* Have histologically confirmed Stage I to III Estrogen Receptor positive (ER+), human epidermal growth factor receptor 2 negative (HER2-) invasive breast carcinoma with Ki-67 >10%
* Be willing and able to provide pre- and on-treatment tumor samples.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Be able to swallow capsules or tablets.
* Be premenopausal women.
* If of childbearing potential must use 1 highly effective method of non-hormonal contraception while receiving study treatment and for the duration specified in protocol.
* Have adequate organ function.

Cohort 2:

* Have a diagnosis of ER+, HER2- early-stage, resected, invasive breast cancer without evidence of distant metastasis
* Have undergone definitive loco-regional therapy.
* Have received at least 5 years of any adjuvant ET.
* Be able to swallow capsules or tablets.
* Be premenopausal women
* Have adequate organ function.
* If of childbearing potential must use 1 highly effective method of non-hormonal contraception while receiving study treatment and for the duration specified in protocol.

Exclusion Criteria:

Cohort 1:

* Have bilateral invasive metastatic.
* occult primary, or inflammatory breast cancer.
* Have had prior bilateral oophorectomy or ovarian ablation.
* Have a serious medical condition
* Had major surgery within 28 days
* Have a history of other cancer (except non melanoma skin cancer, Stage I uterine cancer, or carcinoma in situ of the cervix or other in situ cancer), unless in complete remission with no therapy for a minimum of 1 year.
* Plan to receive concurrent neoadjuvant therapy with any other non-protocol anticancer therapy.
* Have had any prior therapy for an invasive or non-invasive breast cancer.
* Have had prior radiotherapy to the ipsilateral chest wall for any malignancy.
* Have received prior anti-estrogen therapy, including for osteoporosis or prevention of breast cancer.
* Have had prior treatment with any Gonadotropin-releasing hormone (GnRH) agonist within 12 months prior to randomization.
* Receiving current exogenous reproductive hormone therapy

Cohort 2:

* Have presence of ovarian cysts at screening.
* Have metastatic occult primary, or inflammatory breast cancer.
* Have had prior bilateral oophorectomy or ovarian ablation.
* Have a serious medical condition
* Had major surgery within 28 days.
* Have a history of other cancer (except non melanoma skin cancer or carcinoma in situ of the cervix or other in situ cancer), unless in complete remission with no therapy for a minimum of 1 year.
* Completed or discontinued prior adjuvant ET >6 months prior to screening.
* Have received prior therapy with any selective estrogen receptor degrader (SERD).
* Receiving current exogenous reproductive hormone therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Ki-67 Expression | Baseline, Day 29

SECONDARY OUTCOMES:
Change from Baseline in ER Expression | Baseline, Day 29
Change from Baseline in PR Expression | Baseline, Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- United States (5):
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Washington University School of Medicine, St Louis, Missouri
  - Tennessee Oncology, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Oncology Consultants P.A., Houston, Texas
- Belgium (3):
  - Cliniques universitaires Saint-Luc, Brussels
  - Antwerp University Hospital, Edegem
  - UZ Leuven, Leuven
- France (3):
  - CHRU de Brest, Brest
  - Centre de Cancérologie du Grand Montpellier, Montpellier
  - Hôpital Privé Des Côtes d'Armor, Plérin
- Universitaetsklinikum Erlangen, Erlangen, Germany
- Italy (5):
  - Ente Ospedaliero Ospedali Galliera, Genova
  - Humanitas, Milan
  - Humanitas Istituto Clinico Catanese, Misterbianco
  - Nuovo Ospedale di Prato-S.Stefano, Prato
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal should be approved by an independent review panel and researchers should sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Lilly Trials — https://trials.lilly.com/en-US/trial/674818